CLINICAL TRIAL: NCT03103867
Title: Evaluation of Two Different Glucose Monitoring Treatments and Their Impact on Time in Target, Sleep and Quality of Life in Children With Type 1 Diabetes and Primary Caregivers.
Brief Title: QUality of Control and slEep in Children With diabeteS, Using New Technology
Acronym: QUEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Luxembourg (Other)
Responsible Party: Principal Investigator, Carine de Beaufort, Guest Professor , MD, PhD, Centre Hospitalier du Luxembourg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QUEST
Record Dates: First submitted 2017-03-26; First posted 2017-04-06 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CGM augmented pump with PLGS (A) (Experimental): Administration of Subcutaneous administration of Continuous subcutaneous insulin infusion with integrated continuous glucose monitoring and predicted low glucose suspense (PLGS) Randomised cross over treatment during 5 weeks
  Interventions: Device: CGM augmented pump with PLGS ,
- Insulin pump with CGM (B) (Active Comparator): Administration of Subcutaneous administration of Continuous subcutaneous insulin infusion with second device measuring continuous glucose Randomised cross over treatment during 5 weeks
  Interventions: Device: Insulin pump with CGM

INTERVENTIONS:
Device: CGM augmented pump with PLGS , — 5 weeks treatment CGM augmented pump with PLGS compared with 5 weeks treatment with insulin pump with CGM , without integration
  Other Names: 640G, Enlite Sensors , Freestyle Libre
  Arms: CGM augmented pump with PLGS (A)
Device: Insulin pump with CGM — 5 weeks treatment continuous subcutaneous insulin infusion pump with CGM without data integration,
  Other Names: 640G , freestyle libre
  Arms: Insulin pump with CGM (B)

SUMMARY:
The study is an open label single centre randomised cross over study to evaluate the impact of a sensor augmented pump (SAP) with a predictive algorithm to suspend temporarily insulin administration (640G® with the Smart Guard feature) versus the use of the same pump for insulin administration with 'only' continuous glucose measurements (not interacting with the pump, Freestyle Libre ® ) on the time in glucose target , in hypo- and hyperglycemia. Exploratory endpoints are the effect on sleep and quality of life in children with type 1 diabetes and their caregivers.

DETAILED DESCRIPTION:
Optimising metabolic control in children with Type 1Diabetes Mellitus (T1DM) is essential to prevent late complications. Fear of nocturnal hypoglycemia is pervasive amongst parents of children with T1DM, leading to a heightened vigilance by parents to control regularly their children's blood sugar values or to check the sensor information during the night. This leads to chronic sleep interruption and to lack of sleep as well in the parents as in their children with diabetes.

In this study, the impact of new technologies on glucose time in target , hypo fear and quality of life will be evaluated, using continuous interstitial glucose measurements either with a direct impact on insulin administration (640G medtronic pump (R)) and with alerts , or without impact on insulin administration and without alerts.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Duration of diabetes ≥ 6 months
* Insulin pump treatment ≥ 6 months
* HbA1c ≤ 11%
* Parental written informed consent

Exclusion Criteria:

. No parental consent

* Physical or psychological disease likely to interfere with an appropriate conduct of the study
* Current drug therapy knowing to interfere with glucose metabolism
* Chronic sleep medication in the primary caregiver or the patient -

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Time in glucose target | Last 6 days of treatment arm A and last 6 days of treatment arm B
  Percent time in glucose target (3.9 -8 mmol/l) , measured by blinded CGM

SECONDARY OUTCOMES:
time below glucose target | Last 6 days of treatment arm A and last 6 days of treatment arm B
  Percent time spent below glucose target (<3.0mmol/l and < 2,5 mmol/l) measured by blinded CGM (I-Pro 2)
Time above glucose target | Last 6 days of treatment arm A and last 6 days of treatment arm B
  Percent time spent above glucose target (>10.0mmol/l ) measured by blinded CGM (I-Pro 2)
Sleep quantity in patients and caregivers | baselines ( before treatment arm starts) and last week of treatment arm A and last week of treatment arm B
  Total sleep and wake time , number of awakenings measured by wireless actigraph
perception of quality of sleep and quality of life in patients and caregivers | baseline and last week of treatment arm A and last week of treatment arm B
  validated questionnaires
hypoglycaemia fear in patients and caregivers | baseline and last week of treatment arm A and last week of treatment arm B
  Hypoglycemia fear survey for parents and children

CONTACTS AND LOCATIONS:
Overall Officials: Carine de Beaufort, MD,PhD, Study Chair — Centre Hospitalier du Luxembourg
Locations (1):
- Clinique des Enfants CHluxembourg, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schierloh U, Aguayo GA, Fichelle M, De Melo Dias C, Schritz A, Vaillant M, Barnard-Kelly K, Cohen O, Gies I, de Beaufort C. Fear of hypoglycemia and sleep in children with type 1 diabetes and their parents. Front Endocrinol (Lausanne). 2024 Dec 16;15:1419502. doi: 10.3389/fendo.2024.1419502. eCollection 2024. PMID 39736868
- [Derived] Schierloh U, Aguayo GA, Schritz A, Fichelle M, De Melo Dias C, Vaillant MT, Cohen O, Gies I, de Beaufort C. Intermittent Scanning Glucose Monitoring or Predicted Low Suspend Pump Treatment: Does It Impact Time in Glucose Target and Treatment Preference? The QUEST Randomized Crossover Study. Front Endocrinol (Lausanne). 2022 May 31;13:870916. doi: 10.3389/fendo.2022.870916. eCollection 2022. PMID 35712259
- [Derived] Schierloh U, Aguayo GA, Fichelle M, De Melo Dias C, Celebic A, Vaillant M, Barnard K, Cohen O, de Beaufort C. Effect of predicted low suspend pump treatment on improving glycaemic control and quality of sleep in children with type 1 diabetes and their caregivers: the QUEST randomized crossover study. Trials. 2018 Dec 4;19(1):665. doi: 10.1186/s13063-018-3034-4. PMID 30509293